CLINICAL TRIAL: NCT03138382
Title: Effect of Vestibular Stimulation on Fat Consumption and Energy Expenditure as Assessed Using Indirect Calorimetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, V.S. Ramachandran, Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 170798
Record Dates: First submitted 2017-04-25; First posted 2017-05-03 (Actual); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: obesity; metabolic syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: * Crossover design
  * Double-blind
  * Randomized
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment then sham (Experimental): 20 subjects will be randomised to first receive active vestibular nerve stimulation during indirect calorimetry. Then 2 weeks later they will return for sham stimulation during indirect calorimetry.
  Interventions: Device: Vestibular Nerve Stimulator; Device: Sham stimulator
- Sham then treatment (Experimental): 20 subjects will be randomised to first receive sham stimulation during indirect calorimetry. Then 2 weeks later they will return for active vestibular nerve stimulation during indirect calorimetry.
  Interventions: Device: Vestibular Nerve Stimulator; Device: Sham stimulator

INTERVENTIONS:
Device: Vestibular Nerve Stimulator — Electrical stimulation of the vestibular nerve with vestibular nerve stimulator (GVS device) for for 45 minutes using binaural mastoid placement.
Device: Sham stimulator — Looks identical to vestibular nerve stimulator but discharges current into an internal resistor rather than activating the vestibular nerves.

SUMMARY:
There is an ongoing and worsening problem with obesity in the developed, and much of the developing world. Although it has long been realized that Western diets that are rich in sugar and fat play an important role in this, it has only recently been realized that exposure to these diets, particularly in childhood, can damage the part of the brain that determines how much fat there is in the body. The result of this damage is that the so-called "set-point" for fat in this part of the brain is pushed upwards. There is a lot of evidence from animals that activating the brain's balance (vestibular) system pushes this set-point for fat downwards to cause fat loss, probably because this "tricks" the brain into thinking that there is increased physical activity. The aim of this study is to see whether non-invasive electrical stimulation of the vestibular system in human participants causes a change in metabolism of fat and/or energy expenditure, which, if regulated upwards, would suggest this could be used as a means of reducing body fat in humans.

DETAILED DESCRIPTION:
There is a growing realization that obesity can, in many ways, be viewed as a neurological disease triggered by lifestyle factors. There is clear evidence that the central melanocortin system, which is centered in the arcuate nucleus of the hypothalamus, regulates a "set-point" for how much fat the body should have. It does so by altering appetite and metabolic rate so that deviations too far in either direction are strongly resisted. This set-point is determined by genetic, epigenetic and lifestyle factors. Thus, excessive exposure to dietary monosaccharides, such as glucose, and saturated fats, especially in childhood and adolescence, can damage the neurons of the arcuate nucleus and push the set-point up. This then can condemn sufferers to a lifetime of obesity, despite individual efforts to combat it using diet and/or exercise.

Establishing a method of tuning down the set-point for body fat thus has to be a goal if the current obesity pandemic is to be successfully combatted. A significant amount of animal work suggests that stimulating the vestibular system in the inner ear, by means of chronic centrifugation, actually does just that and causes a reduction in body fat. This is likely because chronic vestibular activation is taken by the brain to represent a state of increased physical activity, and in order to optimize homeostasis it would be appropriate for the body to have a leaner physique, by reducing unnecessary energy expenditure from carrying excess fat.

It is possible to stimulate the vestibular nerve in humans by applying a small electrical current to the skin behind the ears. This is an established technology that is believed to be safe, but only previously used for research purposes. The investigators found in a pilot study that recurrent stimulation of this kind for two or three hours a week over four months led to a statistically significant reduction in truncal fat in the active group as opposed to the control group who underwent sham stimulation.

Given the current, and increasing levels of global obesity, it is important to determine whether non-invasive electrical vestibular nerve stimulation (VeNS), otherwise known as galvanic vestibular stimulation (GVS), is a viable treatment option, since if it were this would be of significant scientific importance.

The investigators wish to use the technique of indirect calorimetry to explore this. This involves wearing a tight face mask to collect all inspired oxygen and expired carbon dioxide and using formulae to calculate total energy expenditure and the component of metabolism that is derived from fat as compared to carbohydrate.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Body mass index (BMI) > 25 kg/m2
3. 18-65 years of age inclusive on starting the study.
4. Successfully completed the screening questionnaire.

Exclusion Criteria:

1. History of vestibular dysfunction.
2. History of bariatric surgery, fundoplication, gastric resection or major upper-abdominal surgery (acceptable surgeries include cholecystectomy, hysterectomy).
3. History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears, or of the head and neck.
4. History of weight loss device implantation (e.g. VBloc Maestro or Abiliti).
5. Positive response in Physical Activity Readiness Questionnaire.
6. Currently taking medication for asthma or other breathing conditions.
7. Untreated thyroid disorder (stable treatment for 3 months is acceptable).
8. Other endocrinological causes of weight gain (e.g. Cushing's disease, Cushing's syndrome or acromegaly)
9. Previous diagnosis of HIV infection or AIDS (HIV is known to cause a vestibular neuropathy which would prevent VeNS from working).
10. History of cirrhosis, or liver, kidney or heart failure.
11. Chronic pancreatitis.
12. Treatment with prescription weight-loss drug therapy in the year before starting the study.
13. Tobacco or marijuana smoking in the 6 months prior to study.
14. Known genetic cause of obesity (e.g., Prader-Willi Syndrome).
15. Diabetes mellitus (Types 1 & 2).
16. Diagnosis of epilepsy or use of anti-epileptic medication within six months of starting the study (e.g. for the treatment of peripheral neuropathy)
17. Chronic (more than a month of daily use) treatment with opioid analgesic drugs within the last year.
18. Regular use (more than twice a month) of anti-histamine medication.
19. Use of oral or intravenous corticosteroid medication within two years of starting the study.
20. Use of the beta-blockers atenolol, metoprolol or propranolol within 3 months of starting the study.
21. Current use of tricyclic antidepressant medication for whatever reason.
22. Current alterations in treatment regimens of anti-depressant medication for whatever reason (other than tricyclic antidepressants) (Note: stable treatment regimen for prior six months acceptable).
23. An active diagnosis of cancer.
24. A previous myocardial infarction.
25. A history of stroke or severe head injury (as defined by a head injury that required intensive care). (In case this damaged the neurological pathways involved in vestibular stimulation).
26. Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.).
27. Psychiatric disorders (including untreated severe depression, schizophrenia, substance abuse, bulimia nervosa etc.)
28. Current participant in a clinical trial for weight loss.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Then Sham: 20 subjects will be randomised to first receive active vestibular nerve stimulation during indirect calorimetry. Then 2 weeks later they will return for sham stimulation during indirect calorimetry.
  Vestibular Nerve Stimulator: Electrical stimulation of the vestibular nerve for for 45 minutes using binaural mastoid placement.
  Sham stimulator: Looks identical to vestibular nerve stimulator but discharges current into an internal resistor rather than activating the vestibular nerves.
- Sham Then Treatment: 20 subjects will be randomised to first receive sham stimulation during indirect calorimetry. Then 2 weeks later they will return for active vestibular nerve stimulation during indirect calorimetry.
  Vestibular Nerve Stimulator: Electrical stimulation of the vestibular nerve for for 45 minutes using binaural mastoid placement.
  Sham stimulator: Looks identical to vestibular nerve stimulator but discharges current into an internal resistor rather than activating the vestibular nerves.
Period: Overall Study
Arm/Group | Treatment Then Sham | Sham Then Treatment
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Then Sham: 20 subjects will be randomised to first receive active vestibular nerve stimulation during indirect calorimetry. Then 2 weeks later they will return for sham stimulation during indirect calorimetry.
  Vestibular Nerve Stimulator: Electrical stimulation of the vestibular nerve for for 45 minutes using binaural mastoid placement.
  Sham stimulator: Looks identical to vestibular nerve stimulator but discharges current into an internal resistor rather than activating the vestibular nerves.
- Sham Then Active: 20 subjects will be randomised to first receive sham stimulation during indirect calorimetry. Then 2 weeks later they will return for active vestibular nerve stimulation during indirect calorimetry.
  Vestibular Nerve Stimulator: Electrical stimulation of the vestibular nerve for for 45 minutes using binaural mastoid placement.
  Sham stimulator: Looks identical to vestibular nerve stimulator but discharges current into an internal resistor rather than activating the vestibular nerves.
- Total: Total of all reporting groups
Arm/Group | Active Then Sham | Sham Then Active | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Full Range); unit: years] | 53 [27 to 61] | 47 [34 to 64] | 50 [27 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Fat Consumption (During VeNS)
Description: Change in percent fat utilization from baseline as measured using indirect calorimetry.
Time Frame: During middle 15 minutes of 45 minute vestibular nerve stimulation session
Measure: Mean (Standard Deviation); unit: % of fat as metabolic substrate
Groups:
- Sham: 20 subjects will be randomised to first receive active vestibular nerve stimulation during indirect calorimetry. Then 2 weeks later they will return for sham stimulation during indirect calorimetry.
  Vestibular Nerve Stimulator: Electrical stimulation of the vestibular nerve for for 45 minutes using binaural mastoid placement.
  Sham stimulator: Looks identical to vestibular nerve stimulator but discharges current into an internal resistor rather than activating the vestibular nerves.
- Active: 20 subjects will be randomised to first receive sham stimulation during indirect calorimetry. Then 2 weeks later they will return for active vestibular nerve stimulation during indirect calorimetry.
  Vestibular Nerve Stimulator: Electrical stimulation of the vestibular nerve for for 45 minutes using binaural mastoid placement.
  Sham stimulator: Looks identical to vestibular nerve stimulator but discharges current into an internal resistor rather than activating the vestibular nerves.
Arm/Group | Sham | Active
Number analyzed (Participants) | 20 | 20
% of fat as metabolic substrate | 50.23 (13.05) | 54.44 (14.24)

2. Secondary Outcome: Change in Energy Expenditure (During VeNS)
Description: Change in energy expenditure from baseline in kcal/min as measured using indirect calorimetry.
Time Frame: During middle 15 minutes of 45 minute vestibular nerve stimulation session
Measure: Mean (Standard Deviation); unit: kcal/min
Arm/Group | Sham | Active
Number analyzed (Participants) | 20 | 20
kcal/min | 1.01 (0.26) | 1.02 (0.24)

ADVERSE EVENTS:
Time Frame: During 2 hour period of each both visits.
Description: No adverse events were recorded in this pilot study.
Arm/Group | Treatment Then Sham | Sham Then Treatment
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT03138382/Prot_SAP_000.pdf